CLINICAL TRIAL: NCT04032028
Title: The Thai Red Cross AIDS Research Centre
Brief Title: Same-Day Antiretroviral Therapy Initiation
Status: Active, not recruiting | Type: Observational
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: Same-Day ART Initiation
Record Dates: First submitted 2019-07-02; First posted 2019-07-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Data from a total of 2,500 walk-in or referred individuals who have been confirmed (diagnosed) HIV positive and accessing care and treatment services at the hospitals targeted by this study will be examined. The starting period for this project is estimated to be the last quarter (Q4) of fiscal year 2018.

DETAILED DESCRIPTION:
This 24-month observation study will be conducted in 13 hospitals of 5 provinces in Thailand: Chiang Rai, Chiang Mai, Ubon Ratchathani, Chonburi, and Songkhla. The research team of TRCARC will collect and analyze secondary and de-identified data from the hospitals' databases. In each site, clients who agree to receive Same-Day ART service will go through standard of care procedures at each hospital, which include: post-test counseling and psychosocial support, baseline lab test, clinical screening, and physical examination. The drug regimen prescribed for clients will mirror the first line ART regimen in Thailand's national guideline, which is tenofovir (TDF), emtricitabine (FTC), and efavirenz (EFV). Retention of the clients will reflect that of the hospital's protocol, and CD4 and viral load will be tested according to the national guideline.

ELIGIBILITY:
Inclusion Criteria:

1. Thai nationals
2. HIV-positive status
3. Acceptance of Same-Day ART

Exclusion Criteria:

1. not Acceptance of Same-Day ART

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All persons who have tested HIV positive will be examined.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Acceptance | 5 years
  Acceptance of Same-Day ART
Type of Clients | 5 years
  Type of Clients (newly diagnosed or re-engaged)
Number of clients categorized by demographic characteristics | 5 years
  Demographic Characteristics: age (years), gender (sex at birth and gender identity), risk behavior(s), and reason(s) for HIV testing
Number of clients with each clinical characteristic | 5 years
  Clinical Characteristics based on Thailand's national guidelines (anti-HIV, creatinine, alanine transaminase, syphilis serology, hepatitis B antigen, hepatitis C antibodies, urinalysis, chest X-ray, CD4 count, CDC stage, comorbidity)
Number of clients with each ART drug regimen differ from first line ART regimen | 5 years
  Drug regimen, if different from first line drug (TDF, FTC, EFV)
Duration between date of HIV diagnosis and date of ART initiation | 5 years
  Duration between date of HIV diagnosis and date of ART initiation
Number of clients with each clinical exclusion criteria | 5 years
  Clinical exclusion criterias : suspected TB, suspected cryptococcal meningitis, suspected serious OIs
Duration between date of ART initiation to date of being successfully transferred and date of ART continuation | 5 years
  Duration of linkage to care, if applicable (date of being successfully transferred and date of ART continuation)
Retention | 5 years
  Retention (retention in care, discontinued ART, loss to follow-up, death) at month 1, month 3, month 6, and month 12 after ART initiation
Viral load count | 5 years
  Viral load count (VL tested, percentage of VL suppressed, and dates of VL suppressed)

CONTACTS AND LOCATIONS:
Locations (11):
- Thailand (11):
  - Thai Red Cross AIDS Research Centre, Pathum Wan, Bangkok
  - Wat Yannasangwararam Hospital, Bang Lamung, Changwat Chon Buri
  - Queen Savang Vadhana Memorial Hospital, Chon Buri, Changwat Chon Buri
  - Sunpasitthiprasong Hospital, Udon Thani, Changwat Ubon Ratchathani
  - Hangdon Hospital, Hang Dong, Chiang Mai
  - Nakornping Hospital, Mae Rim, Chiang Mai
  - Sarapee Hospital, Saraphi, Chiang Mai
  - Hat Yai Hospital, Hat Yai, Song Khla
  - Sanpatong Hospital, Chiang Mai
  - Chiang Mai Hospital, Chiang Mai
  - Chiang rai prachanukor Hospital, Chiang Rai

REFERENCES:
- [Derived] Seekaew P, Phanuphak N, Teeratakulpisarn N, Amatavete S, Lujintanon S, Teeratakulpisarn S, Pankam T, Nampaisan O, Jomja P, Prabjunteuk C, Plodgratoke P, Ramautarsing R, Phanuphak P. Same-day antiretroviral therapy initiation hub model at the Thai Red Cross Anonymous Clinic in Bangkok, Thailand: an observational cohort study. J Int AIDS Soc. 2021 Dec;24(12):e25869. doi: 10.1002/jia2.25869. PMID 34967504